CLINICAL TRIAL: NCT03831152
Title: A Phase 3B Open-Label Extension Of Study B23CS (ARENA 2) Evaluating The Continued Safety And Efficacy Of ADV7103 In Subjects With Primary Distal Renal Tubular Acidosis
Brief Title: Extension Study in Primary Distal Renal Tubular Acidosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients enrolled. Study no longer required due to completion of long term safety study in the EU.
Sponsor: Advicenne Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B24CS
Record Dates: First submitted 2019-01-23; First posted 2019-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acidosis, Renal Tubular
MeSH Terms: conditions — Acidosis, Renal Tubular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental ADV7103 (Experimental): All patients receive ADV7103 at their individualized dose
  Interventions: Drug: ADV7103

INTERVENTIONS:
Drug: ADV7103 — Single group assignment

SUMMARY:
Open-label study involving longitudinal assessment of the continued safety, tolerability, and efficacy of ADV7103 in maintaining targeted serum bicarbonate levels, preventing metabolic acidosis, and preventing hypokalemia in the following groups of subjects with primary dRTA:

1. subjects who participated in Study B23CS and were adherent to the protocol;
2. subjects ≥ 6 months of age who are living in Europe and did not participate in Study B23CS; and
3. infants younger than 6 months of age

ELIGIBILITY:
Inclusion Criteria:

Subjects who participated in Study B23CS must meet all of the following criteria to be registered into this study:

1. Female or male subjects who participated in Study B23CS and were adherent to the protocol;

Subjects who did not participate in Study B23CS must meet all of the following criteria to be registered into this study:

1. Female or male subjects ≤ 65 years of age at time of consent with the following stipulations:

   1. Subjects ≥ 6 months of age must reside in Europe
   2. Subjects < 6 months of age must reside in the United States, Canada, or Europe;
2. Subjects < 6 months of age must be able to swallow (not suck) solid food without difficulty;
3. Subject presents with a previous diagnosis of primary dRTA;
4. Subject ≥ 6 months of age requires ≥ 0.9 mEq/kg/day of alkali therapy to maintain serum bicarbonate levels above the LLN;
5. Urine pH > 5.5 and serum bicarbonate > 18 mEq/L for subjects ≥ 4 years old or > 17 mEq/L for subjects < 4 years old on alkali therapy and potassium supplementation (if indicated) on at least one occasion for each within 6 months;
6. European subjects must be included in a social health insurance system and/or in compliance with the recommendations of the national law in force relating to biomedical research;
7. Subject or parent/guardian is willing and able to understand and sign informed consent and willing to comply with protocol instructions; child assent when appropriate; and

Exclusion Criteria:

Subjects who participated in Study B23CS and meet any of the following criteria will be considered ineligible for registration into this study:

1. Female subject who is pregnant or lactating or has plans for pregnancy during the study; or
2. Subject requires therapy with potassium sparing diuretics, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, trimethoprim, drospirenone and other progestins, nephrotoxic antibiotics, penicillins, tacrolimus, or medications known to delay gastric emptying or otherwise interfere with absorption of study product.

Subjects who did not participate in Study B23CS and meet any of the following criteria will be considered ineligible for registration into this study:

1. Female subject who is pregnant or lactating or has plans for pregnancy during the study;
2. Subject has evidence of proximal tubule dysfunction unless the subject is < 6 months of age;
3. Subject presents with another diagnosed condition as a potential etiology for her/his dRTA ;
4. Subject requires therapy with potassium sparing diuretics, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, trimethoprim, drospirenone and other progestins, nephrotoxic antibiotics, penicillins, tacrolimus, or medications known to delay gastric emptying or otherwise interfere with absorption of study product;
5. Subject has evidence of obstructive uropathy or other findings on renal ultrasound expected to require intervention during the course of the study;
6. Subject has any of the following laboratory abnormalities:

   1. AST and/or ALT > 1.5x upper limit of normal (ULN)
   2. Serum potassium > 5.0 mEq/L or hypokalemia accompanied by clinical symptoms (eg, muscle cramps) or significant ECG changes (eg, T wave depression, U wave elevation)
   3. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (according to the updated Schwartz formula for children and Chronic Kidney Disease - Epidemiology Collaboration [CKD-EPI] formula for adults)
   4. Total bilirubin > ULN, except with known Gilbert's disease.
7. Subject has been hospitalized or had outpatient surgery (other than minor skin and dRTA disease-related procedures or ear tube placement) in the past 6 months or is planning surgery in the next 6 months.

Ages: 4 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The Safety of ADV7103 will be assessed by evaluating the frequency of Treatment-Emergent Adverse events as compared to placebo | To 30 months
  Number/proportion of subjects presenting with ADV7103 treatment-related adverse events (AEs) during the study, by severity grade.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Ulmann, M.D., Ph.D., Study Chair — Advicenne Pharma
Locations (1):
- University of South Florida Pediatric Infectious Diseases, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No